CLINICAL TRIAL: NCT02111382
Title: Electroencephalography Activity in Individuals With Nonspecific Chronic Low Back Pain After Cranial Osteopathic Manipulative Treatment: Study Protocol of a Randomized, Controlled Crossover Trial
Brief Title: Electroencephalography Activity in Individuals With Nonspecific Chronic Low Back Pain After Cranial Osteopathic Manipulative Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The pilot study demonsttated some new concerns about methodology. So we decided to suspended temporarily to added new settings to study design.
Sponsor: University of Brasilia (Other)
Collaborators: University Hospital of Brasília (Unknown)
Responsible Party: Principal Investigator, Wagner Rodrigues Martins, Professor, PhD, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: cv4-2014
Record Dates: First submitted 2014-03-28; First posted 2014-04-11 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2018-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; osteopathic manipulations; electroencephalography
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CV4 (4th ventricle technique) technique (Experimental): Will be conduced a real cranial osteopathic medicine technique.
  Interventions: Other: CV4 Cranial (4th ventricle technique) Osteopathic Manipulative
- CV4 sham (Sham Comparator): This group will received only a sham manual therapy technique.
  Interventions: Other: CV4 (4th ventricle technique) manual therapy sham technique
- Control (No Intervention): The participants will be in supine position for 5 minutes without any visual or verbal contact.

INTERVENTIONS:
Other: CV4 Cranial (4th ventricle technique) Osteopathic Manipulative — The participant will be in supine position during the whole procedure. The practitioner sits behind the participant's head, contacts participant's lateral protuberances of the squama occipitalis (medially to the occipitomastoid suture) with the thenar eminence of both hands.
  When the practitioner feels the PRM (a pulsating rhythm caused by liquor production and reabsorption), the flexion phase will be resisted and the extension phase exaggerated. The compressive force is held until the PRM stops (event known as 'Still point'). The compression will be held until the practitioner feels PRM gradual return; the compression will be slowly diminished, and then, the practitioner remove the hands from the occipital bone, laying the participant's head on the table.
  The CV4 technique will be performed by an osteopath D.O. - member of the Brazilian Register of Osteopaths.
  Other Names: 4th ventricle technique
  Arms: CV4 (4th ventricle technique) technique
Other: CV4 (4th ventricle technique) manual therapy sham technique — The participant will be in supine position and the practitioner will be seated behind the participant's head. The practitioner places the fingers (2nd to 5th) under the occipital bone, touching only the squama occipitalis. The practitioner will hold this position for 5 minutes, and after this period the participant's head will be placed on the table.
  The CV4 sham will be performed by a registered physiotherapist.
  Arms: CV4 sham

SUMMARY:
Osteopathic medicine is based on a diagnostic and therapeutic system to treat tissue mobility/ motility dysfunctions in general, using different approaches (depending on the target tissue) known as osteopathic manipulative treatment.

Among all the available techniques those ones addressed to the cranial field are most questioned because of the lack of scientific evidence; but the compression of the 4th ventricle technique has been largely studied in clinical trials. Studies have shown that the technique may affect both central and autonomous nervous system, modulating some reflexes (Traube-Hering baro signal), and modifying brain cortex electrical activity through central sensitization in subjects with chronic low back pain.

Thus, investigators hypothesize that the compression of the 4th ventricle may modulate peak alpha frequency (electroencephalographic assessment) and promote physical relaxation in subjects in vigil.

DETAILED DESCRIPTION:
A randomized controlled crossover trial with blinded assessor was designed to test the hypothesis. A total of 81 participants will be assigned to three treatment conditions, with seven days of washout: compression of the 4th ventricle group; sham compression of the 4th ventricle group; control group (no intervention).

All participants will be recruited at the Outpatient Rehabilitation Service of the University Hospital of Brasília - University of Brasília (Brazil).

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old with self-reported nonspecific chronic low back pain will be recruited

Exclusion Criteria:

* Participants suffering from secondary chronic low back pain,
* fever, chills, sweating, weight loss, asthenia, anorexia;
* cardiovascular and respiratory symptoms such as chest pain, dyspnea and cough;
* headache, dizziness, lightheadedness, fainting, tremors, dysarthria and aphasia;
* participants who underwent surgery on the spine;
* diagnosis of any neurological, cardiac, respiratory and rheumatic disease;
* regular use of drugs with effects on the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Peak alpha frequency (Electroencephalography) | Baseline, 10 minutes.
  Baseline: before intervention. 10 minutes: 10 minutes after intervention.

SECONDARY OUTCOMES:
Pain intensity | Baseline, 10 minutes
  Baseline: before intervention. 10 minutes: 10 minutes after intervention. Pain intensity: 0-10 Numeric Pain Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wagner Martins, PhD, Principal Investigator — Assistant Professor, PhD - Graduate Program in Physical Therapy Universidade de Brasília (UnB) - Faculdade de Ceilândia (FCE)
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Jakel A, von Hauenschild P. Therapeutic effects of cranial osteopathic manipulative medicine: a systematic review. J Am Osteopath Assoc. 2011 Dec;111(12):685-93. PMID 22182954
- [Background] Licciardone JC, Brimhall AK, King LN. Osteopathic manipulative treatment for low back pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2005 Aug 4;6:43. doi: 10.1186/1471-2474-6-43. PMID 16080794
- [Background] Nelson KE, Sergueef N, Lipinski CM, Chapman AR, Glonek T. Cranial rhythmic impulse related to the Traube-Hering-Mayer oscillation: comparing laser-Doppler flowmetry and palpation. J Am Osteopath Assoc. 2001 Mar;101(3):163-73. PMID 11329812
- [Background] Shi X, Rehrer S, Prajapati P, Stoll ST, Gamber RG, Downey HF. Effect of cranial osteopathic manipulative medicine on cerebral tissue oxygenation. J Am Osteopath Assoc. 2011 Dec;111(12):660-6. PMID 22182951
- [Background] Huneke NT, Brown CA, Burford E, Watson A, Trujillo-Barreto NJ, El-Deredy W, Jones AK. Experimental placebo analgesia changes resting-state alpha oscillations. PLoS One. 2013 Oct 11;8(10):e78278. doi: 10.1371/journal.pone.0078278. eCollection 2013. PMID 24147129
- [Background] Field T, Diego M, Hernandez-Reif M. Tai chi/yoga effects on anxiety, heartrate, EEG and math computations. Complement Ther Clin Pract. 2010 Nov;16(4):235-8. doi: 10.1016/j.ctcp.2010.05.014. Epub 2010 Jun 29. PMID 20920810
- [Background] Cutler MJ, Holland BS, Stupski BA, Gamber RG, Smith ML. Cranial manipulation can alter sleep latency and sympathetic nerve activity in humans: a pilot study. J Altern Complement Med. 2005 Feb;11(1):103-8. doi: 10.1089/acm.2005.11.103. PMID 15750368
- [Background] Miana L, Bastos VH, Machado S, Arias-Carrion O, Nardi AE, Almeida L, Ribeiro P, Machado D, King H, Silva JG. Changes in alpha band activity associated with application of the compression of fourth ventricular (CV-4) osteopathic procedure: a qEEG pilot study. J Bodyw Mov Ther. 2013 Jul;17(3):291-6. doi: 10.1016/j.jbmt.2012.10.002. Epub 2012 Nov 16. PMID 23768271
- [Background] Jensen MP, Gertz KJ, Kupper AE, Braden AL, Howe JD, Hakimian S, Sherlin LH. Steps toward developing an EEG biofeedback treatment for chronic pain. Appl Psychophysiol Biofeedback. 2013 Jun;38(2):101-8. doi: 10.1007/s10484-013-9214-9. PMID 23532434
- [Background] Klem GH, Luders HO, Jasper HH, Elger C. The ten-twenty electrode system of the International Federation. The International Federation of Clinical Neurophysiology. Electroencephalogr Clin Neurophysiol Suppl. 1999;52:3-6. No abstract available. PMID 10590970
- [Derived] Martins WR, Diniz LR, Blasczyk JC, Lagoa KF, Thomaz S, Rodrigues ME, de Oliveira RJ, Bonini-Rocha AC. Immediate changes in electroencephalography activity in individuals with nonspecific chronic low back pain after cranial osteopathic manipulative treatment: study protocol of a randomized, controlled crossover trial. BMC Complement Altern Med. 2015 Jul 13;15:223. doi: 10.1186/s12906-015-0732-2. PMID 26165865
- See also: University of Brasilia — http://www.unb.br
- See also: Brazilian Register of Osteopaths — http://www.registrodososteopatas.com.br